CLINICAL TRIAL: NCT02600169
Title: Retrospective Analysis of Response Markers and Adverse Events in a Nationwide Cohort of Advanced Melanoma Patients Treated With Pembrolizumab
Brief Title: Retrospective Analysis of Response Markers and Adverse Events in Melanoma Patients Treated With Pembrolizumab
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 20150907
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with pemprolizumab: All patients in this study have received treatment with pembrolizumab for the indication of an advanced melanoma. Patients will be included from all 14 WIN-O (Werkgroep Immunologie Nederland voor Oncologie) centers in the Netherlands. Patients are at least 18 years of age.
  Interventions: Drug: Pemprolizumab

INTERVENTIONS:
Drug: Pemprolizumab — All patients in this study have received treatment with pembrolizumab for the indication of an advanced melanoma.
  Other Names: MK3475

SUMMARY:
This study is a retrospective cohort study. A database will be created from the data available of all patients that have participate in the named patient program for pembrolizumab in the Netherlands. This database will be used for analysis of response markers and for an evaluation of adverse events.

DETAILED DESCRIPTION:
This study is a retrospective cohort study. A database will be created from the data available of all patients that have participate in the named patient program for pembrolizumab in the Netherlands. This database will be used for analysis of response markers and for an evaluation of adverse events.

ELIGIBILITY:
All patients that were eligible for treatment with pembrolizumab in the Named Patient Program in the Netherlands.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study have received treatment with pembrolizumab for the indication of an advanced melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Early serum response markers | up to day 126
  Serum markers: S100B, LDH, white blood count differential neutrophils, monocytes, lymphocytes, eosinophils, basophils. Markers will be correlated to early response as measured by RECIST 1.1 criteria at week 12 and 18 of treatment with pembrolizumab.
Predicitve patient characteristics | baseline
  Patient characteristics: age, gender, WHO performance status
Predictive tumor characteristics | baseline
  Tumor characteristics: M-stage, presence of CNS metastases, mutation status, PD-L1 status.
Adverse events of clinical interest will be collected and graded according to the CTCAE version 4.0 criteria | 2 years

SECONDARY OUTCOMES:
Survival | 2 years
  Overall survival will be evaluated for all patients treated with pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: G.A.P. Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands